CLINICAL TRIAL: NCT00904384
Title: Prevalencia, Factores de Riesgo y características patogénicas Diferenciales de EPOC y Enfisema en Pacientes Con infección VIH.
Brief Title: Prevalence and Determinants of Chronic Obstructive Pulmonary Disease (COPD) in HIV+ Patients
Acronym: HIV&COPD
Status: Completed | Type: Observational
Sponsor: Cimera (Network)
Collaborators: Hospital Universitari Son Dureta (Other)
Responsible Party: Dr Melchor RIERA JAUME, Hospital Universitario Son Dureta
Other Study IDs: IB956/08 IP
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: HIV Infections; COPD
Keywords: HIV+; COPD; emphysema
MeSH Terms: conditions — HIV Infections; Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV+: Patients with HIV infection living in the Autonomous Community of the Balearic Islands (CAIB), Spain
- Reference group: Same determinations as in HIV+ cases will be obtained in the control group of COPD patients without HIV infection as part of the study PAC-EPOC (FIS 05/2082)

SUMMARY:
The prevalence of COPD in HIV+ and AIDS patients is unknown. The pathophysiology of HIV infection and COPD might be of interest to both conditions. The research hypotheses of this study are:

In patients with HIV infection living in the Autonomous Community of the Balearic Islands (CAIB):

1. The Prevalence of airflow obstruction in patients with HIV infection is higher than in the general population.
2. In these patients, the prevalence of emphysema detected by HRCT is common (greater than or equal to 15%)
3. DLCO measurement is a good marker for the presence of emphysema on CT
4. The inflammatory response is different from that seen in patients with COPD and / or emphysema without HIV infection

DETAILED DESCRIPTION:
Objectives

Main objective To determine the prevalence of COPD

Secondary objectives

1. To determine the prevalence (and severity) of emphysema (HRCT)
2. To Identify risk factors associated with the development of COPD and / or emphysema
3. To analyze the predictive value of measuring DLCO as a marker of emphysema by HRCT
4. To determine the prevalence of lung function abnormalities deeming specific drug treatment (bronchodilators, inhaled corticosteroids) in the absence of clinical symptoms
5. To compare the pattern of inflammatory response in patients with COPD and / or emphysema, with and without HIV infection

Methodology:

Cross-sectional, descriptive, study of up to 350 patients with HIV infection.

All the patients will be be assessed with:

1. an standardized clinical questionnaire
2. full lung function tests
3. high resolution CT scan
4. induced sputum for bacterial culture, P. jiroveci, proinflamatory citokines (cytokines array)
5. blood analysis: hemogram; basic biochemistry; HIV predictors; autoantibodies; proinflammatory citokines (ultrasensitive ELISA); C reactive protein (ultrasensitive nephelometry)
6. exhaled gases (NO and CO)

Statistical analysis:

Description of the univariate distribution of the categorical or ordinal variables will be realized with a table of frequencies, and in quantitative variables by means of measures of central tendency (mean or median) and dispersion (standard deviation or 95 % confidence intervals). Depending on the normality of the distribution of variables, any comparisons will be assessed by means of parametric tests (T test; Chi2) or non parametric tests (Mann Whitney). To explore relationships between the variables of study, Kolgomorov-Smirnov for the comparison of groups and analysis of regression bivariate, and multivariate (logistic regression), will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection in stable phase (minimum of three months)
* Being followed-up in external HUSD consultations (on a regular basis)
* Age 40-69 years

Exclusion Criteria:

* Chronic non-respiratory disease in terminal stage (stage IV or V of chronic kidney failure, heart failure, advanced chronic liver disease (Child C))
* Lack of cooperation
* Estimated survival of less than 1 year or Karnofsky <70
* Pregnancy
* Opportunistic infection in the last month
* Post lung resection
* Systemic treatment with corticosteroids, immunosuppressive chemotherapy or interferon at the time of inclusion

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the HIV outpatient consultation of the Internal Medicine Department of Hospital Universitario Son Dureta (HUSD), in Mallorca, Spain. The HUSD is the tertiary, reference hospital in the CAIB.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2008-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of airflow obstruction compatible with COPD in patients with HIV infection | cross-sectional

SECONDARY OUTCOMES:
To determine the prevalence (and severity) of emphysema (HRCT) | Cross-sectional
To Identify risk factors associated with the development of COPD and / or emphysema | Cross-sectional
To analyze the predictive value of measuring DLCO as a marker of emphysema by HRCT | Cross-sectional
To determine the prevalence of lung function abnormalities deeming specific drug treatment (bronchodilators, inhaled corticosteroids) in the absence of clinical symptoms | Cross-sectional
To compare the pattern of inflammatory response in patients with COPD and / or emphysema, with and without HIV infection | Cross-sectional

CONTACTS AND LOCATIONS:
Overall Officials: Melchor Riera, MD, Principal Investigator — Hospital Universitario Son Dureta
Locations (1):
- Hospital Universitario Son Dureta, Palma de Mallorca, Balearic Islands, Spain

REFERENCES:
- See also: Hospital Universitario Son Dureta — http://www.hsd.es